CLINICAL TRIAL: NCT05019573
Title: A Double-blind Placebo Controlled Study to Determine the Effect of Tea Consumption on Gut Microbiota Composition and Body-Iron Status
Brief Title: Can the Reduction of Iron Availability Caused by Tea Consumption Change the Gut Microbiota Composition and Disrupt Host Body-iron Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Gemma Walton, Principle Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: UREC 20/04
Record Dates: First submitted 2021-06-15; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Focus of Study: 1- Effect of Tea Consumption on Gut Microbiota; Focus of Study: 2- Effect of Tea Consumption on Body-iron Status
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind (subject/investigator), placebo controlled, parallel study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black tea group (Experimental): Volunteers meeting inclusion/exclusion criteria will be given an appropriate number of black tea samples twice a day with main meals for the 4 weeks of the treatment.
  Interventions: Dietary Supplement: Black tea
- Placebo group (Placebo Comparator): Volunteers meeting inclusion/exclusion criteria will be given an appropriate number of placebo tea samples twice a day with main meals for the 4 weeks of the treatment.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Black tea — Black tea twice a day for 4 weeks
  Arms: Black tea group
Dietary Supplement: Placebo — Placebo tea twice a day for 4 weeks
  Arms: Placebo group

SUMMARY:
Iron is an essential micronutrient for nearly all living organisms, including microbes. The adult human body contains approximately 3-5 g of iron (45-55 mg/kg of body weight in adult women and men, respectively). Iron-deficiency related anaemia (IDA) is a major public health problem that affects more than 2 billion people globally and this represents 24.8% of the world's population. According to World Health Organisation (WHO), iron deficiency is the most common cause of anaemia worldwide, with infants, children and women at higher risk, making it a global public health problem. Much iron deficiency is a result of poor iron dietary absorption since iron is poorly absorbed (~15%). Absorption inhibition factors (iron chelators) like phytate and tannins, found in tea and vegetables have been reported to act as potent iron uptake inhibitors. Despite its health benefits, tea-containing polyphenols (tannins) have been associated with reduction and disruption of iron absorption, acting as inhibitors of non-haem iron uptake, potentially resulting in poor iron status. However, most studies on the effect of tea on iron absorption are largely based on isotope-labelled single meal studies and animal studies. Iron is a requirement of many microorganisms, as such changes in iron availability can also have an impact on the gut microbiota. Long-term controlled human intervention studies to investigate the effect of tea on iron absorption and the effect on gut microbiota composition are scarce. In addition, the impact of dietary tannins on the gut microbiota is not understood. Thus, this proposed human intervention trial will investigate the combined effect of tea-tannins on iron status, inflammation and gut microbiota composition. This will be the first study to consider this combination of factors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* Gender: Male or Female
* Volunteers agree to sign an informal written consent form
* General good health
* Normal haemoglobin and serum ferritin levels

Exclusion Criteria:

* Regular tea drinkers
* Use of antibiotics, prebiotics or probiotics (in food products or as supplements), laxatives, anti-spasmodic, anti-diarrhoea drugs, (e.g. Orlistat, Lactulose) in the last 4 weeks prior to, or during the study period.
* Use of any iron supplement in the last 6 months prior to the study period.
* If participants have received bowel preparation for investigative procedures in the 4 weeks prior to the study.
* Surgical resection of any part of the bowel.
* If you have any chronic gut disorder/disease, such as IBS, IBD, etc. or other conditions that might affect the gut environment, e.g. coeliac disease. If participants are taking any medication that could affect the iron absorption (e.g. lansoprazole, omeprazole). Those with gluten allergies (e.g. Celiac disease) must be excluded as the placebo may contain gluten
* If participants are pregnant or are lactating.
* If participants have a BMI > 30 kg/m2.
* Severe allergy or any history of severe abnormal drug reaction, drug or alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Composition and diversity of the faecal microbiota of the individuals consuming tea/placebo during the 4 weeks intervention | 4 weeks intervention
  Changes in composition and diversity of faecal microbiota in response to black tea intervention assessed by next generation sequences NGS
Levels of faecal and urine metabolites of the individuals consuming tea/placebo during the 4 weeks intervention | 4 weeks intervention
  Changes of metabolic profile during the intervention will be estimated in faecal and urine samples using Nuclear Magnetic Resonance (NMR)
Levels of ferritin (ng/mL) as body-iron status indicators of the individuals consuming tea/placebo during the 4 weeks intervention | 4 weeks intervention
  Ferritin will be monitored through blood samples collected during study visits.
Changes in the concentration (pg/mL) of inflammation markers in plasma of the individuals consuming tea/placebo using enzyme-linked immunosorbent assays (ELISAs) | 4 weeks intervention
  gut inflammation will be assessed by measuring concentration (pg/mL) of gut inflammatory markers as plasma intestinal fatty acid-binding protein and cytokines from plasma (e.g. IL-10, IL-6, TNFα). Samples will be analysed using enzyme-linked immunosorbent assays (ELISAs)
Changes in the concentration (mcg/g) of faecal calprotectin (gut inflammatory marker) during tea intervention using enzyme-linked immunosorbent assays (ELISAs) | 4 weeks intervention
  Gut inflammation will be assessed measuring concentration (mcg/g) of calprotectin. Increase in the levels of Calprotectin indicates the migration of neutrophils to the intestinal mucosa, which occurs during intestinal inflammation.

SECONDARY OUTCOMES:
Assessment of stool consistency | 4 weeks intervention
  The Bristol stool chart will be provided to volunteer to measure stool consistency, the chart rate the stool consistency from 1-7 (solid - liquid) based on the shape of stool.
Assessment of gastrointestinal symptoms | 4 weeks intervention
  Daily assessment of gastrointestinal symptoms (abdominal pain, bloating or flatulence) will be recorded daily using daily diary.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF